CLINICAL TRIAL: NCT06660043
Title: Influence of Bodily Practices on the Quality of Life of Women
Brief Title: Influence of Bodily Practices on the Quality of Life of Women With Endometriosis
Acronym: PCKendo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 665-PCKendo
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- physical activity (Experimental)
  Interventions: Other: physical activity
- analgesic physical therapy (Active Comparator)
  Interventions: Other: analgesic physical therapy
- analgesic physical therapy AND physical activity (Experimental)
  Interventions: Other: analgesic physical therapy AND physical activity

INTERVENTIONS:
Other: physical activity — 40 min circuit training session
  Arms: physical activity
Other: analgesic physical therapy — physical therapy with massage and Transcutaneous Electrical Nerve Stimulation in a 40min session
  Arms: analgesic physical therapy
Other: analgesic physical therapy AND physical activity — 25 min circuit training session and 15 min physical therapy
  Arms: analgesic physical therapy AND physical activity

SUMMARY:
This research focuses on understanding how physical activity can improve the quality of life for women with endometriosis by enhancing their self-perception, particularly regarding their physical abilities and appearance. The study is based on the idea that improving internal perceptions can lead to better overall well-being for these women. Previous studies, suggest that physical self-perception plays a crucial role in shaping an individual's quality of life. There is also evidence supporting a reciprocal relationship between physical self-concept and participation in physical activity

In this context, the research aims to explore how physical activity could positively influence the self-concept of women suffering from endometriosis, which in turn could enhance their quality of life. By focusing on improving both physical abilities and body image through regular exercise, this study seeks to offer insights into potential therapeutic approaches for managing the physical and psychological impacts of endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Menstruating women aged 18 to 55;
* proven diagnosis of endometriosis (pelvic ultrasound or MRI)
* Having endometriosis-related pain of a level higher than 3 on the VAS scale and/or chronic incapacitating symptoms related to endometriosis;
* Patient without treatment or with stable endometriosis treatment (pill and/or ATG) who has not undergone treatment during the last 6 months;
* Patient affiliated to a health insurance scheme;
* French-speaking patient;
* Patient having given free, informed and express oral consent.

Exclusion Criteria:

* Any patient whose endometriosis treatment has been modified for less than 6 months;
* Having endometriosis-related pain greater than or equal to 8 on the VAS scale;
* Cardiovascular risks related to physical training;
* Inability to perform proposed exercises;
* Patient under guardianship;
* Patient deprived of liberty;

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of quality of life | 6months
  EHP-30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Frederique PERROTTE, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Physical Therapy Studio, Chevry-Cossigny
  - Hôpital Saint Joseph, Paris

IPD SHARING:
Plan to Share IPD: No